CLINICAL TRIAL: NCT02242396
Title: A Study of a Hypertensive Population Under Treatment With Micardis® and Micardis Plus® Under Real Clinical Conditions With the Goal to Control the Early Morning BP Rise (SURGE II)
Brief Title: A Study of a Hypertensive Population Under Treatment With Micardis® and Micardis Plus® to Control the Early Morning BP Rise (SURGE II)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.496
Record Dates: First submitted 2014-09-16; First posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; telmisartan, hydrochlorothiazide drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hypertensive patients
  Interventions: Drug: Telmisartan; Drug: Telmisartan hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis®
Drug: Telmisartan hydrochlorothiazide
  Other Names: Micardis Plus®

SUMMARY:
The primary objective was to evaluate, through the use of Home blood pressure monitoring (HBPM), the degree of BP control in the early morning hours after 8 weeks of treatment in patients with essential hypertension under treatment with Micardis®, Telmisartan or Micardis Plus®, Telmisartan hydrochlorothiazide.

The co-primary endpoints were the degree of BP control, and change from baseline until study end in mean systolic blood pressure (mSBP) and mean diastolic blood pressure (mDBP) HBPM in the early morning hours after 8 weeks of treatment with Micardis®, Telmisartan or Micardis Plus®, Telmisartan hydrochlorothiazide.

Secondary endpoints were office BP control rates, office BP response rates, and reduction in mSBP and mDBP Office blood pressure measurement (OBPM) from baseline to final visit, discontinuations and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Patients male or female between 18 and 80 years of age
* Patients with mild to moderate essential hypertension
* Patients diagnosed with hypertension that are not currently taking antihypertensive medication or previously diagnosed hypertensive patients who are uncontrolled with their current treatment

Exclusion Criteria:

* Pre-menopausal women who have no birth control, who are pregnant or nursing
* Patients with advanced hepatic impairment or advanced renal impairment
* Patients with New York Heart Association (NYHA) functional class III or IV congestive heart failure (CHF), unstable angina, acute myocardial infarction, heart surgery or stroke within the previous six months
* Patients with any type of relevant arrhythmia according to the assessment of the investigator
* Patients with any valvular disease with hemodynamic repercussion
* Patients receiving chronic administration of oral anticoagulants or digoxin
* Patients with known hypersensitivity to any component in the formulation of Micardis®, Telmisartan or Micardis Plus®, Telmisartan hydrochlorothiazide
* Patients with previous history of angioedema associated with angiotensin converting enzyme (ACE) inhibitors
* Patients with severe, uncontrolled hypertension or any form of secondary hypertension
* Patients with any other clinical conditions which, in the opinion of the investigator, would not allow for the safe completion of the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive population under real life clinical practice in an ambulatory setting
Sampling Method: Non-Probability Sample
Enrollment: 5248 (Actual)
Dates: Start 2005-08; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Change of degree of Blood Pressure (BP) control in the early morning hours | 8 weeks of treatment
Change from baseline in mSBP and mDBP by HBPM in the early morning | Baseline, after 8 weeks of treatment
  BP control during the morning time-periods (6:00 to 11:59), BP < 135/85 mmHg (HBPM: mean of morning measurements)

SECONDARY OUTCOMES:
Change from baseline in office BP control rates | Baseline, after 8 weeks
Change from baseline in office BP response rates | Baseline, after 8 weeks
Reduction in mSBP and mDBP by OBPM | Baseline, after 8 weeks
Number of patients with adverse events | up to 8 weeks
Global Assessment of tolerability by investigator on a 6-point scale | after 8 weeks
Global assessment efficacy by investigator on 6-point scale | after 8 weeks